CLINICAL TRIAL: NCT05440227
Title: A Phase II, Double Blind, Randomized, Placebo-controlled Study of PG2 Injection for the Treatment of moderate-to Severe Fatigue in Patients With Locally Advanced, Recurrent, or Metastatic Breast Cancer Who Are Receiving Infusional Chemotherapy
Brief Title: PG2 Injection for the Treatment of moderate-to Severe Fatigue in Breast Cancer Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: PhytoHealth Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PH-CP032
Record Dates: First submitted 2022-06-27; First posted 2022-06-30 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Cancer-related Fatigue
Keywords: breast cancer; fatigue; CRF
MeSH Terms: conditions — Breast Neoplasms; Fatigue | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PG2 treatment group (Experimental): 500 mg PG2 injection will be administered to this group once per week for 8 weeks.
  Interventions: Drug: PG2 Lyo. Injection 500mg
- Placebo-controlled group (Experimental): Placebo injection will be administered to this group once per week for 8 weeks.
  Interventions: Drug: Placebo 0.9% normal saline

INTERVENTIONS:
Drug: PG2 Lyo. Injection 500mg — PG2 Lyo. Injection 500mg (reconstituted with 0.9% normal saline 500ml) will be administered weekly for 8 weeks.
  Arms: PG2 treatment group
Drug: Placebo 0.9% normal saline — 0.9% normal saline 500ml will be administered weekly for 8 weeks.
  Arms: Placebo-controlled group

SUMMARY:
The objective of this study is to assess the efficacy of weekly PG2 regimen as a complementary treatment for patients with recurrent unresectable (local or regional) or metastatic breast cancer who experienced moderate to severe fatigue while receiving chemotherapies.

DETAILED DESCRIPTION:
The objective of this study is to assess the efficacy of weekly PG2 regimen as a complementary treatment for patients with recurrent unresectable (local or regional) or metastatic breast cancer who experienced moderate to severe fatigue while receiving chemotherapies. The primary endpoint is to examine whether PG2, compar ed with placebo, can successfully reduce patients' fatigue (observed via prorated area under the curve [AUC] for the Brief Fatigue Inventory [BFI] scores) when primed with PG2 for 8 weeks during their chemotherapy. The other efficacy endpoints including th e time course change of patient reported BFI, fatigue improvement response rate (fatigue improvement response is defined as those with at least 10% reduction from baseline in the total BFI scores) after 8 weeks, self perceived improvement, hematological improvement, health related quality of life, and safety profiles will also be assessed between treatment arms and compared with the baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged ≥ 20 years
2. ECOG performance score ≤ 2
3. Locally advanced, recurrent or metastatic, histologically documented breast cancer who is currently undergoing infusional chemotherapy regimen.
4. Presence of moderate to severe cancer related fatigue prior to randomization as defined by at least two records of usual fatigue score ≥ 4 on the numeric scale (0 -10), which must be ≥ 14 days apart.
5. Laboratory values obtained prior to randomization:

   * Hgb ≥ 10 g/dL (patients must not be transfused ≤ 14 days to meet this criterion)
   * Creatinine ≤ 1.2 x ULN
   * AST (SGOT) or ALT (SGPT) ≤1.5 x ULN (or ≤5.0 x ULN for patients with liver metastases)
6. Pain under controlled of score ≤ 4 on the numeric scale (0 -10)
7. Life expectancy ≥ 3 months
8. Ability to complete patient questionnaires alone or with assistance.
9. Negative pregnancy test done ≤ 14 days prior to randomization, for women of childbearing potential only, and willing to take efficient contraceptives procedures to avoid pregnancy throughout the study period.
10. Willing to provide written informed consent and agree to follow the study requirements.

Exclusion Criteria:

1. Known brain metastasis or primary CNS malignancy
2. Has known psychiatric or substance abuse disorders.
3. Malnutrition, active infection, uncontrolled thyroid disorder, uncontrollable hypertension or diabetes mellitus, significant pulmonary disease and cardiovascular disease.
4. Currently using any other pharmacologic agents.
5. Subject who is unwilling to receive transfusions when, at the investigator's discretion, it is required to control her anemia.
6. Other medical conditions that necessitate chronic systemic use of steroids (e.g. use of prednisolone > 10 mg daily or equivalent steroids fore more than 2 weeks).
7. ≤ 4 weeks from major surgery to randomization, including any procedure that requires general anesthetics.
8. Pain requiring opioid pain medication, however, over the counter analgesics such as acetaminophen or ibuprofen are allowed.
9. Use of monoamine oxidase inhibitors (MAOI) (such as Moclobemide).
10. Planning to start or complete any type of cancer therapy during the 8 weeks course of the study, once randomized on the study.
11. Use of any over the counter herbal/dietary supplement marketed for fatigue or energy.
12. Known history of hypersensitivity to Astragalus products.
13. Currently participating another interventional study or planning to join one in the upcoming 8 weeks after randomization.
14. Currently breast feeding.
15. With any other serious disease considered by the investigator not in the condition to enter into the trial.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-05-17 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Prorated AUC for the global BFI score | 8 weeks
  The prorated AUC for the global BFI score (average scores of 9 items), usual fatigue (item2) and worst fatigue (item 3) will be compared between PG2 and the placebo arms at the end of the study.

SECONDARY OUTCOMES:
Fatigue improvement response rate (FIRR) | 8 weeks
  FIRR is defined as those with at least 10% reduction from baseline in the total BFI scores after 8-week treatment. 20% and 30% reduction will also be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Wu Chen, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No